CLINICAL TRIAL: NCT01511380
Title: Targeting HIV Risk Behaviors in Juvenile Drug Court-Involved Youth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA025880 (NIH)
Record Dates: First submitted 2012-01-04; First posted 2012-01-18 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2013-05

CONDITIONS: Substance Use; Sexual Risk Behaviors
Keywords: juvenile; randomized trial; substance abuse; sexual risk; contingency management
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risk Reduction Therapy for Adolescents (Experimental): Youth randomly assigned to RRTA will complete a family focused treatment program that will work with the youth and his or her caregiver to help reduce youth substance use and risky sexual behavior using principals of behavior modification and contingency management.
  Interventions: Behavioral: Risk Reduction Therapy for Adolescents
- Usual services (Active Comparator): For youth randomly assigned to usual treatment services, the youth will receive the treatment services recommended by the drug court.
  Interventions: Behavioral: Usual services

INTERVENTIONS:
Behavioral: Risk Reduction Therapy for Adolescents — This project integrates CM and a family systems intervention for sexual risk with evidence-based family engagement strategies, and tests this intervention in a juvenile drug court setting. Due to the individualized nature of the proposed intervention, the specific course of treatment will vary by youth and family. Based on our experience with clinic-based treatment models it is anticipated that most families will remain in active treatment for 4-6 months and that, during this time, they will attend approximately 1-2 sessions per week, for 1-2 hours per session.
  Arms: Risk Reduction Therapy for Adolescents
Behavioral: Usual services — In addition to the standard juvenile drug court requirements, youth randomly assigned to the usual services condition are also ordered to receive treatment services from the local state or privately-funded alcohol and drug treatment provider agencies. The service delivery model for agencies typically includes intensive outpatient, traditional outpatient, and home-based services, depending upon assessment of youth and family needs. Groups focus on risk reduction, peer influence, conflict resolution, and anger management. Additionally, youth might receive treatment pertaining to drug selling behavior, individual sessions and/or family group therapy. The theoretical orientations of the provider agencies are cognitive-behavioral and systems theory. Interventions are not usually manual driven, and selection of material is typically left to the therapists' discretion.
  Arms: Usual services

SUMMARY:
This study is designed to gain knowledge about effective interventions for reducing HIV risk in a high risk population. A new Risk Reduction Therapy for Adolescents (RRTA) will be compared to usual services received by youth in juvenile drug courts. It is expected that youth treated with RRTA will show greater reductions in substance use and risky sexual behaviors. Reducing HIV risk by effectively targeting substance use and risky sexual behaviors in high-risk groups such as juvenile drug court-involved youth could favorably impact society at multiple levels (individual, family, peer, community, fiscal).

DETAILED DESCRIPTION:
The overriding purpose of this study is to develop and test an intervention for reducing substance use and risky sexual behaviors among youth involved in juvenile drug court. Juvenile drug court provides an excellent setting in which to pursue the key study objectives by providing access to a well identified high risk population. Second, in addition to frequent judicial oversight, juvenile drug courts include several features that can enhance intervention effectiveness, sustainability, and potential for adoption. In addition, the fact that all juvenile drug courts have community-based treatment components and that such courts have been disseminated nationwide suggests the possibility of eventual widespread adoption if the proposed intervention is effective. The proposed intervention integrates evidence-based protocols for contingency management (CM) for substance abusing youth and family engagement strategies, with an evidence-informed family systems intervention for sexual risk originally developed to address substance use and sexual risk behaviors in HIV+ youth. These three interventions will be integrated into an efficient intervention that, if effective, can be amenable to adoption by juvenile drug courts. Following protocol development and beta testing, 160 drug court youth and their families will be randomized to the experimental intervention condition (Risk Reduction Therapy for Adolescents or "RRTA") versus Drug Court with Community Services (DC) conditions. Key outcomes will be assessed through 18-months post-baseline using a multi-method approach that will include assessment of substance use, risky sexual behaviors, criminal behavior, and participation in HIV counseling and testing services. Specific aims include: 1: Adapt existing intervention and training protocols into a single, efficient RRTA intervention, beta test this RRTA protocol with four youth in juvenile drug court and their families, and revise treatment and research protocols accordingly; 2: Conduct a randomized trial with 160 youth in juvenile drug court and their families to examine youth-level intervention effects (i.e., on substance use, sexual risk behavior, HIV counseling and testing, delinquent behavior) in comparison to DC through 18- months post referral and assess intervention fidelity. 3. If results suggest a positive RRTA treatment effect, revise the intervention and training protocols in preparation for an effectiveness study and extended follow-up study. Importantly, the proposed study will (1) consider the multiple levels of influence on juvenile drug use, criminal justice involvement, and HIV risk behaviors, (2) integrate a drug abuse and HIV prevention intervention for youth in the criminal justice system with drug-related offenses, (3) address health disparities by targeting a primarily minority population of youth, and (4) increase referrals to HIV testing and counseling of drug court-involved youth. This study is designed to reduce HIV risk by addressing the potent interaction of drug use and risky sexual behaviors in drug court youth with evidence-based treatment components to maximize the likelihood of reversing these youths' adverse behavioral trajectories.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in juvenile drug court or pre-enrollment status
* residing with permanent caregiver
* youth and caregiver fluent in English

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in substance use frequency | Baseline through 18 months post-baseline
  Self-reported substance use by the adolescent will be assessed using a variation of the Form 90. Urine drug screens for cannabis, cocaine, opiates, methamphetamines, and amphetamines will be collected using the "5-Test Integrated Cup" supplied by BioTechNostix.

SECONDARY OUTCOMES:
Change in delinquent behavior | Baseline through 18 months post-baseline
  The 47-item Self-Report Delinquency Scale will be used to tap violent offending, general delinquency, and status offenses. Archival records maintained by state juvenile justice authorities will be used to examine youths' involvement in the juvenile and adult justice systems.
Change in sexual risk behaviors | Baseline through 18 months post-baseline
  The measure of sexual risk behaviors was selected to maximize the likelihood of identifying the highest-risk sexual behaviors. The Sexual Risk Behavior Scale has been used in previous HIV studies. This measure will be used to assess participant sexual encounters over the past 3 months and condom use during vaginal and anal sex.
Change in frequency of HIV counseling and testing | Baseline through 18 months post-baseline
  Participation in HIV counseling and testing will be assessed using a standardized set of questionnaire items. Baseline questions will assess participants' lifetime history of voluntary HIV counseling and testing and identical questions will be re-administered at 6, 12 and 18 months post-baseline to assess whether youth received HIV counseling and testing at any point since the baseline interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States